CLINICAL TRIAL: NCT00645671
Title: A Randomized Multicenter, Double-Masked, Parallel-Group Clinical Safety and Efficacy Evaluation of Loteprednol Etabonate Ophthalmic Ointment, 0.5% Versus Vehicle for the Treatment of Inflammation Following Cataract Surgery
Brief Title: Loteprednol Etabonate Ophthalmic Ointment vs. Vehicle in the Treatment of Inflammation Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 525
Record Dates: First submitted 2008-03-13; First posted 2008-03-28 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Ocular Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol Etabonate (Experimental): Loteprednol etabonate 0.5% ophthalmic ointment
  Interventions: Drug: 0.5% Loteprednol Etabonate Ophthalmic Ointment
- Vehicle (Placebo Comparator): Vehicle of loteprednol etabonate ointment
  Interventions: Drug: Vehicle of Loteprednol Etabonate Ophthalmic Ointment

INTERVENTIONS:
Drug: 0.5% Loteprednol Etabonate Ophthalmic Ointment — 1/2 inch ribbon four times a day for 14 days
  Arms: Loteprednol Etabonate
Drug: Vehicle of Loteprednol Etabonate Ophthalmic Ointment — 1/2 inch ribbon four times a day for 14 days
  Arms: Vehicle

SUMMARY:
To evaluate the clinical safety and efficacy of Loteprednol Etabonate Ophthalmic Ointment, 0.5% vs. vehicle for the treatment of inflammation following cataract surgery

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are candidate for routine, uncomplicated cataract surgery
2. Subjects who, in the Investigator's opinion, have potential postoperative pinholed Snellen visual acuity (VA) of at least 20/200 in the study eye.

Exclusion Criteria:

1. Subjects who will require concurrent ocular therapy with NSAIDs, mast cell stabilizers, antihistamines, decongestants, or immunosuppressants (e.g., Restasis), or with ocular or systemic corticosteroids
2. Subjects who have known hypersensitivity or contraindication to the study drug(s) or their components
3. Subjects who are monocular or have pinholed Snellen VA 20/200 or worse in the non-study eye
4. Subjects who have had ocular surgery (including laser surgery) in the study eye within 3 months or in the fellow eye within 2 weeks prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyson J Berliner, MD/PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- John Hunkeler, MD, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 400 subjects, 18 years old or older who were candidates for routine, uncomplicated cataract surgery, were enrolled at 17 investigative sites in the US. First subject was enrolled on 3/14/2008 and last subject visit was 3/23/2009.
Pre-assignment Details: Following cataract surgery at visit 3 (post operative day 1), subjects were assessed for eligibility. 201 subjects were randomized to receive loteprednol etabonate ointment and 199 to receive its vehicle.
Period: Overall Study
Arm/Group | Loteprednol Etabonate | Vehicle
Started | 201 | 199
Completed | 200 | 193
Not Completed | 1 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate | Vehicle | Total
Number analyzed (Participants) | 201 | 199 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.39) | 69.2 (8.77) | 69.2 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 119 | 237
  Male | 83 | 80 | 163
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 6 | 7
  Black or African American | 17 | 12 | 29
  White | 183 | 179 | 362
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Complete Resolution of Anterior Chamber Cells and Flare. Grade=0.
Description: A combination of the grades for inflammatory cells and flare in the anterior chamber. Cells: accumulation of white blood cells in aqueous. 0=No cells seen; 1=1-5 cells; 2=6-15 cells; 3=16-30 cells; 4= >30 cells. Flare: Scattering of a slit lamp light beam when directed into the anterior chamber (Tyndall effect). 0=None; 1=Mild; 2=Moderate; 3=Severe; 4=Very severe.
Time Frame: Postoperative Day 8 (Visit 5)
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 201 | 199
participants
  Yes | 48 | 27
  No | 153 | 172

2. Secondary Outcome: Subjects With Complete Resolution of Anterior Chamber Cells and Flare. At Each Follow-up Visit.
Description: as for outcome 1
Time Frame: At each follow-up visit through day18 (Visit 7)
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 201 | 199
participants
  Visit 4 (postoperative day 3) | 10 | 9
  Visit 5 (postoperative day 8) | 48 | 27
  Visit 6 (postoperative day 15) | 84 | 30
  Visit 7 (postoperative day 18) | 86 | 39

3. Secondary Outcome: Change From Baseline to Each Follow-up Visit in Anterior Chamber Cells and Flare
Description: as for outcome 1
Time Frame: Baseline and each follow-up visit through day18 (Visit 7)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Composit scores
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 201 | 199
Composit scores
  Visit 4 (postoperative day 3) | -1.0 (1.08) | -0.4 (1.42)
  Visit 5 (postoperative day 8) | -2.1 (1.31) | -0.7 (1.81)
  Visit 6 (postoperative day 15) | -2.6 (1.37) | -0.9 (1.97)
  Visit 7 (postoperative day 18) | -2.5 (1.45) | -1.1 (1.95)

4. Primary Outcome: Grade 0 for Pain
Description: Pain: A positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching. Grade 0 = None; 1=Minimal; 2=Mild; 3=Moderate; 4=Moderately Severe; 5=Severe
Time Frame: Postoperative Day 8 (Visit 5)
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 201 | 199
participants
  Yes | 156 | 90
  No | 45 | 109

ADVERSE EVENTS:
Time Frame: The LE treatment group had a mean exposure of 13.2 days (+/-3.06), the vehicle treatment group mean exposure was 9.2 days (+/-5.10). Mean days of exposure was < 14 days due to the use of rescue medication, especially in the vehicle group.
Description: Ocular AE's in study eyes and were reported prior to rescue medication use - safety population.
Arm/Group | Loteprednol Etabonate | Vehicle
Serious Adverse Events (participants affected / at risk) | 3/201 | 2/199
Other Adverse Events (participants affected / at risk) | 110/201 | 161/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=201) | Vehicle (N=199)
Endophthalmitis (Eye disorders) | 1 (1) | 1 (1) — Unrelated to study drug but related to the cataract surgery.
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Unrelated to study drug and study participation, associated with an accidental injury.
Myocardial Infarction (Cardiac disorders) | 1 (2) | 1 (2) — unrelated to study drug and study participation, due to a concurrent condition
Post-operative inflammation (Eye disorders) | 1 (1) | 1 (1) — Corneal Macular Edema, possibley related to study drug, probably related to study participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=201) | Vehicle (N=199)
Anterior chamber cell (Eye disorders) | 5 (15) | 10 (15)
Anterior chamber inflammation (Eye disorders) | 61 (167) | 106 (167)
Ciliary hyperemia (Eye disorders) | 5 (15) | 10 (15)
Conjunctival hyperemia (Eye disorders) | 10 (25) | 15 (25)
Corneal edema (Eye disorders) | 8 (19) | 11 (19)
Eye pain (Eye disorders) | 8 (34) | 26 (34)
Iritis (Eye disorders) | 11 (30) | 19 (30)
Lacrimation increased (Eye disorders) | 6 (20) | 14 (20)
Ocular hyperemia (Eye disorders) | 5 (15) | 10 (15)
Ocular pruritis (Eye disorders) | 5 (21) | 16 (21)
Photophobia (Eye disorders) | 17 (36) | 19 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with, the Sponsor and such that confidential or proprietary information is not disclosed.

Prior to publication or presentation, a copy of the final text should be forwarded by the Investigator(s) to the Sponsor or its designee for comment.